CLINICAL TRIAL: NCT02028442
Title: A Clinical Study Of Enadenotucirev Administered by Sub-Acute Fractionated Intravenous Injection: Dose Escalation in Metastatic Epithelial Solid Tumours and Randomised Controlled Trial in Metastatic Colorectal Cancer
Brief Title: Phase I / II Study of Enadenotucirev by Sub-acute Fractionated IV Dosing in Cancer Patients
Acronym: EVOLVE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ColoAd1-1001
Record Dates: First submitted 2013-10-29; First posted 2014-01-07 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Solid Tumours of Epithelial Origin; Metastatic Colorectal Cancer; Metastatic Bladder Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Urinary Bladder Neoplasms | interventions — enadenotucirev

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enadenotucirev (Experimental)
  Interventions: Biological: Enadenotucirev

INTERVENTIONS:
Biological: Enadenotucirev — Oncolytic virus

SUMMARY:
This is a multicentre, open-label, Phase I/II study of enadenotucirev in patients with either solid tumour of epithelial origin not responding to standard therapy or for whom no standard treatment exists (Phase I dose escalation stage Single cycle), mCRC not responding to standard therapy (Phase I dose escalation Repeat cycle cohort expansion stage ), mCRC not responding to standard therapy or advanced or metastatic bladder cancer not candidate for chemotherapy (Phase Ib) or mCRC in stable disease or partial response after 3-4 months of first line standard of care chemotherapy (Phase II).

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent
* Age ≥ 18 years and the patient must be at least the legal age limit to be able to give consent within the jurisdiction the study is taking place.
* ECOG performance status 0 or 1
* Predicted life expectancy of 3 months or more
* Ability to comply with study procedures in the Investigator's opinion
* Recovered to Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies
* Adequate renal function

  * Creatinine ≤ 1.5 mg/dL or calculated creatinine clearance using the Cockcroft-Gault formula ≥ 60 mL/min, or measured creatinine clearance ≥ 60 mL/min, Haematuria: dipstick ≤ 2+
  * Proteinuria: dipstick ≤ 2+
* Adequate hepatic function

  * Serum bilirubin < 1.5 mg/dL
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3x upper limit of normal (ULN)
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Haemoglobin ≥ 100 g/L for UCC and ≥ 90 g/L for other cancers
* Adequate coagulation tests: international normalised ratio (INR) ≤ 1.5 x ULN
* For females of childbearing potential (defined as <2 years after last menstruation or not surgically sterile), a negative serum pregnancy test must be documented within 14 days prior to first administration of study treatment
* For women who are not postmenopausal (24 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use two adequate methods of contraception, during the treatment period and for at least 3 months after the last dose of study drug
* For men: agreement to use a barrier method of contraception during the treatment period and for at least 6 months after the last dose of study drug
* At least 3 weeks since any dose of IV systemic chemotherapy and at least two weeks since any oral dose of capecitabine at the time of first administration of ColoAd1.

Phase I Specific Inclusion Criteria:

Dose Escalation Stage only (except Repeat Cycle Cohort):

- Solid tumour of epithelial origin not responding to standard therapy or for whom no standard treatment exists

Dose Expansion Stage Single Cycle and Dose Escalation Stage Repeat Cycle Cohort:

* mCRC not responding to standard therapy
* ≤ 3 prior lines of systemic therapy for advanced disease OR ≤ 4 prior lines of systemic therapy for advanced disease if one of the 4 lines was an anti EGFR therapy given as a single agent or combined to a previously administered chemotherapy regimen Phase Ib:mCRC not responding to standard therapy
* no more than 3 prior lines of systemic therapy for advanced disease OR no more than 4 prior lines of systemic therapy for advanced disease if one of the 4 lines was an anti EGFR therapy given as a single agent or combined to a previously administered chemotherapy regimen
* Advanced or metastatic UCC, who have received a maximum of one chemotherapy-containing regimen and a maximum of one other systemic treatment with biologic agents only.

Phase II Specific Inclusion Criteria:

* mCRC
* Have received 3 - 4 months of first line chemotherapy with either FOLFOX, FOLFIRI or CAPOX, with or without bevacizumab
* At least one measurable lesion according to RECIST 1.1 criteria
* Documented partial response or stable disease
* Eligible to receive chemotherapy with FOLFOX or CAPOX after a short chemotherapy interruption (3 to 4 weeks)

Exclusion Criteria for all Patients:

* Pregnant or breast feeding females;
* Known history or evidence of significant immunodeficiency due to underlying illness (e.g. human immunodeficiency virus [HIV]/acquired immunodeficiency syndrome [AIDS]) and/or medication (e.g. systemic corticosteroids, or other immunosuppressive medications including cyclosporine, azathioprine, interferons, within the past 4 weeks)
* Splenectomy
* Prior allogeneic or autologous bone marrow or organ transplantation
* Active infections requiring antibiotics, physician monitoring, or recurrent fevers >38.0 degrees centigrade associated with a clinical diagnosis of active infection
* Active viral disease or known positive serology for HIV, hepatitis B or hepatitis C;
* Use of the following anti-viral agents: ribavirin, adefovir, lamivudine or cidofovir within 7 days prior to day 1; or pegylated interferon (PEG-IFN) (within 14 days prior to first administration of ColoAd1)
* Administration of an investigational drug within 28 days prior to first dose of ColoAd1
* Major surgery within 4 weeks or radiotherapy within 3 weeks prior to first dose of ColoAd1
* Another primary malignancy within the past 3 years (except for non melanoma skin cancer or cervical cancer in situ)
* Central nervous system (CNS) metastasis that is symptomatic and/or requires treatment
* Any condition or illness that, in the opinion of the Investigator or the medical monitor, would compromise patient safety or interfere with the evaluation of the safety of the drug
* Known allergy to treatment medication or its excipients
* Any other medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent

Phase II Specific Exclusion Criteria:

* Progression on first line therapy
* A complete response on first line therapy
* Use of first line therapy for longer than 4 months
* Use of any first line treatment with a chemotherapy regimen other than FOLFOX, FOLFIRI or CAPOX (each with or without bevacizumab)
* More than 6 weeks since the last administration of 5 FU, capecitabine, oxaliplatin or irinotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-09-20 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2016-04-29 (Actual)

PRIMARY OUTCOMES:
Phase 1 - Maximum Tolerated Dose | Up to Day 22
  - Maximum tolerated dose (MTD) / maximum feasible dose (MFD) of enadenotucirev when administered by sub-acute fractionated IV injection (phase I Dose Escalation) and recommended dose for phase II.
Phase 1b - Selection of suitable schedule for repeat cycle IV administration | Up to Day 134
  Open label assessment of 2 repeat cycle schedules, with expansion cohort at the MTD or MFD with best repeat cycle schedule in advanced/metastatic UBC patients.

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (3):
  - GZA ziekenhuizen campus Sint-Augustinus, Wilrijk, Antwerp
  - Cliniques Universitaires St Luc, Brussels
  - Ghent University Hospital, Ghent
- Spain (3):
  - Institut Catala d Oncologica, Barcelona
  - START - Hospital Universitario Madrid Sanchinarrio, Madrid
  - Hospital Universitario Virgen del Rocio (HUVR), Seville

REFERENCES:
- [Derived] Khalil DN, Prieto Gonzalez-Albo I, Rosen L, Lillie T, Stacey A, Parfitt L, Soff GA. A tumor-selective adenoviral vector platform induces transient antiphospholipid antibodies, without increased risk of thrombosis, in phase 1 clinical studies. Invest New Drugs. 2023 Apr;41(2):317-323. doi: 10.1007/s10637-023-01345-8. Epub 2023 Mar 10. PMID 36897458
- [Derived] Machiels JP, Salazar R, Rottey S, Duran I, Dirix L, Geboes K, Wilkinson-Blanc C, Pover G, Alvis S, Champion B, Fisher K, McElwaine-Johnn H, Beadle J, Calvo E. A phase 1 dose escalation study of the oncolytic adenovirus enadenotucirev, administered intravenously to patients with epithelial solid tumors (EVOLVE). J Immunother Cancer. 2019 Jan 28;7(1):20. doi: 10.1186/s40425-019-0510-7. PMID 30691536
- See also: Journal publication for EVOLVE study — https://jitc.bmj.com/content/7/1/20